CLINICAL TRIAL: NCT01561703
Title: Postoperative Healthcare Utilization in Adenotonsillectomy Patients With Postoperative Antibiotic Administration Compared to Patients Without Antibiotic Administration
Brief Title: Comparing Healthcare Utilization Between Adenotonsillectomy Patients With and Without Postoperative Antibiotic Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200310
Record Dates: First submitted 2012-03-16; First posted 2012-03-23 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-11

CONDITIONS: Snoring; Strep Throat
Keywords: Healthcare utilization; Tonsillectomy; Adenoidectomy/Tonsillectomy; Antibiotics
MeSH Terms: conditions — Snoring | interventions — Anti-Bacterial Agents; Amoxicillin; Clavulanic Acid; Amoxicillin-Potassium Clavulanate Combination; Azithromycin; Cefaclor; Cephalexin; Cefdinir; Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anitibiotic (Experimental): Patients will receive postoperative antibiotic after surgery.
  Interventions: Drug: Antibiotic
- Control (No Intervention): Patients will NOT receive postoperative antibiotic

INTERVENTIONS:
Drug: Antibiotic — One of seven antibiotics (amoxicillin; amoxicillin/clavulanate potassium; azithromycin; cefaclor; cephalexin; cefdinir; or clindamycin) will be given at standard dosage that may be used for 7-10 days following surgery .
  Other Names: Amoxicillin; Amoxicillin/ and clavulanate potassium/Augmentin; Azithromycin/Zithromax; Cefaclor/Ceclor; Cephalexin; Cefdinir/Omnicef; Clindamycin/Cleocin Pediatric
  Arms: Anitibiotic

SUMMARY:
This study is designed to look at healthcare utilization following the removal of tonsils and adenoids in pediatric patients who are not given an antibiotic following surgery.

DETAILED DESCRIPTION:
The objective for this trial is to provide evidence that not prescribing postoperative antibiotics increases the number of phone calls to the physician, increases the number of emergency department/urgent care/clinic visits in the postoperative period, and increases medical diagnostic costs (ie: labwork, cultures, x-rays). Additionally, the investigators aim to provide evidence that a higher percentage of patients not given a prescription for antibiotics will ultimately obtain a prescription from another provider.

One of the most common surgical procedures performed in the pediatric population is tonsillectomy. The term "tonsillectomy" refers to the surgical excision of the entire tonsil tissue and may or may not include excision of the adenoid tissue as well. Typical symptoms following surgery are pain, malaise, and fever among others. Otolaryngologists for many years have prescribed antibiotics postoperatively based on early randomized controlled trials that suggested a benefit in improved recovery. A recent poll showed that 79% of otolaryngologists routinely prescribe antibiotics to reduce postoperative morbidity and not for antibiotic prophylaxis. The American Academy of Otolaryngology-Head and Neck Surgery (AAOHNSF) recently published an evidenced-based Clinical Practice Guideline for tonsillectomy in children in which the routine use of postoperative antibiotics was evaluated. Evaluation of more recent literature showed that routine use of post-operative antibiotics does not show benefit in improving the main measures of perioperative morbidity . Multiple individual trials showed that antibiotic use had no impact on pain, amount of analgesic use, recovery time, or time required to return to a normal diet. However, routine antibiotic use for prevention of postoperative fever remains in controversy and has shown benefit in two trials and while showing no benefit in two different trials. Considering the lack of supporting evidence of benefit in reducing postoperative morbidity, the AAOHNSF has issued a strong recommendation against the routine administration of postoperative antibiotics for tonsillectomy.

The investigators experience as a very busy pediatric surgical service is that in the 1-2 weeks following tonsillectomy, physicians and clinics commonly receive phone calls from concerned parents regarding local and referred pain, bad breath, and fever. Despite patient education at several steps during the process, parental phone calls regarding postoperative fever remain common. While post-operative fever is known to occur following tonsillectomy, management of this issue on the phone, sometimes over the weekend, can be challenging. Children are often in pain, more tired than usual, and not eating well. Even though these are all anticipated symptoms, when they occur with fever, it is difficult to provide adequate reassurance to a concerned parent. Often parents think their child has an infection and are expecting that their provider will start an antibiotic. From the clinician perspective, it can be difficult to discern whether or not there is a concurrent illness that should be evaluated. As a result, parents often bring their children to an urgent care clinic, emergency department, or physician clinic for evaluation and may eventually obtain an antibiotic prescription for their complaints to cover a possible infection.

While routine use of antibiotics does not show benefit in improving many of the main elements of morbidity, controversy remains regarding reduction of postoperative fever. When a fever occurs in a child who is not taking an antibiotic, parents often become concerned about an infection and desire an antibiotic and further evaluation. The concern of the parent in some cases leads to unnecessary visits to emergency departments, urgent care clinics, and physician clinics for evaluation. The workup performed in the evaluation of these patients may include complete blood count, chest x-ray, urinalysis, and urine cultures. Ultimately, the patient may be given an empiric antibiotic prescription. To date there has been no literature documenting healthcare utilization compared between patients who were given antibiotics and those who were not given antibiotics. The goal of this study is to evaluate healthcare utilization and patient/caregiver burden between these groups. If increased healthcare utilization and patient/caregiver burden is found in the "no antibiotic" group, then analysis of the type of utilization and outcome will direct future efforts to improve patient education regarding postoperative morbidity or possibly to continue routinely administering post operative empiric antibiotics. This will benefit in the effort to improve patient satisfaction with surgery, reduce unnecessary healthcare costs, and reduce unnecessary antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for Adenotonsillectomy or Tonsillectomy only (AT/T).
* Patient age 18 years or younger(if patient not 18 years, then parent/guardian will be the participant and must also meet inclusion criteria #3).
* English as the primary language.

Exclusion Criteria:

* Patients not having English as their primary language
* Patients <18 years of age without a parent/guardian present.
* Patients with periodic fever syndrome, immunocompromise, hemophilia, cerebral palsy, down syndrome, sickle cell disease, or with known preoperative aspiration.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliav Gov-Arie, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Background] Telian SA, Handler SD, Fleisher GR, Baranak CC, Wetmore RF, Potsic WP. The effect of antibiotic therapy on recovery after tonsillectomy in children. A controlled study. Arch Otolaryngol Head Neck Surg. 1986 Jun;112(6):610-5. doi: 10.1001/archotol.1986.03780060022002. PMID 3516177
- [Background] Colreavy MP, Nanan D, Benamer M, Donnelly M, Blaney AW, O'Dwyer TP, Cafferkey M. Antibiotic prophylaxis post-tonsillectomy: is it of benefit? Int J Pediatr Otorhinolaryngol. 1999 Oct 15;50(1):15-22. doi: 10.1016/s0165-5876(99)00228-1. PMID 10596882
- [Background] Krishna P, LaPage MJ, Hughes LF, Lin SY. Current practice patterns in tonsillectomy and perioperative care. Int J Pediatr Otorhinolaryngol. 2004 Jun;68(6):779-84. doi: 10.1016/j.ijporl.2004.01.010. PMID 15126019
- [Background] Baugh RF, Archer SM, Mitchell RB, Rosenfeld RM, Amin R, Burns JJ, Darrow DH, Giordano T, Litman RS, Li KK, Mannix ME, Schwartz RH, Setzen G, Wald ER, Wall E, Sandberg G, Patel MM; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: tonsillectomy in children. Otolaryngol Head Neck Surg. 2011 Jan;144(1 Suppl):S1-30. doi: 10.1177/0194599810389949. PMID 21493257

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Patients will receive postoperative antibiotic after surgery.
  Amoxicillin: Generic antibiotic at standard dosage that may be used for 7-10 days following surgery .
  Amoxicillin/clavulanate potassium: Generic antibiotic given at standard dosage that may be used for 7-10 day after surgery
  Azithromycin: Generic antibiotic given at standard dosage that may be used for 7-10 day after surgery
  Cefaclor: Generic antibiotic given at standard dosage that may be used for 7-10 day after surgery
  Cephalexin: Generic antibiotic given at standard dosage that may be used for 7-10 day after surgery
  Cefdinir: Generic antibiotic given at standard dosage that may be used for 7-10 day after surgery
  Clindamycin: Generic antibiotic given at standard dosage that may be used for 7-10 day after surgery
- Control: Patients will NOT receive postoperative antibiotic
  No postoperative antibiotic: Patients will not be given a prescription for postoperative antibiotics
Period: Overall Study
Arm/Group | Intervention | Control
Started | 28 | 30
Completed | 20 | 24
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 20 | 24 | 44
Age, Customized [Number; unit: participants]
  <18 years | 20 | 24 | 44
Gender [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Healthcare Utilization
Description: Questionnaire designed to evaluate healthcare utilization following surgery. Unit of measure will be the number of participants utilizing each category of healthcare.
Time Frame: 6 wks post-operative appointment
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 20 | 24
participants
  Reported Fever | 5 | 16
  Made a phone call to clinic | 5 | 8
  ER/UR/Clinic visit | 2 | 9
  Received "additional" antibiotic | 0 | 6
  Diagnostic workup at ER | 0 | 6

ADVERSE EVENTS:
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/24
Other Adverse Events (participants affected / at risk) | 0/20 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes